CLINICAL TRIAL: NCT02135380
Title: A Prospective, Multicentric, Phase I/II, Open Label, Randomized, Interventional Study to Evaluate the Safety and Efficacy of Intravenous Autologous Adipose Derived Adult Stem Cells for Treatment of Idiopathic Pulmonary Fibrosis (IPF).
Brief Title: Evaluate Safety and Efficacy of Intravenous Autologous ADMSc for Treatment of Idiopathic Pulmonary Fibrosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasiak Research Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KRPL/IPF/11-12/002
Record Dates: First submitted 2014-05-08; First posted 2014-05-09 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Autologous Stromal Vascular Fraction (Other): Single dose of autologous adipose derived Stromal Vascular Fraction (SVF) intravenously.
  Interventions: Biological: Autologous Stromal Vascular Fraction (SVF)
- Autologous Adipose Derived MSCs (Other): 3 doses of 2 million per kg body weight adipose tissue derived Ex-vivo expanded Mesenchymal stem cells (MSC) intravenously each. All the three doses will be given at weekly intervals.
  Interventions: Biological: Autologous Adipose Derived MSCs (ADMSCs)
- Control (Active Comparator): * corticosteroids i.e. Prednisolone ≤10mg/day or ≤20 mg every alternate day
  * Immunosuppressants like Cyclophosphamide or Azathioprine at a dose of 2mg/kg/day not exceeding 150 mg/day
  * Antioxidants like N-acetylcysteine (NAC) at a dose upto 1800 mg/day.
  * Pirfenidone at dose upto 1200 to 1800 mg/day
  Interventions: Other: Control

INTERVENTIONS:
Biological: Autologous Stromal Vascular Fraction (SVF) — Study arm A subjects will receive single dose of autologous adipose derived Stromal Vascular Fraction (SVF) intravenously.
  Other Names: Autologous Stromal Vascular Fraction
  Arms: Autologous Stromal Vascular Fraction
Biological: Autologous Adipose Derived MSCs (ADMSCs) — Study arm B subjects will receive total 3 doses of 2 million per kg body weight adipose tissue derived Ex-vivo expanded Mesenchymal stem cells (MSC) intravenously each. All the three doses will be given at weekly intervals.
  Other Names: Autologous Adipose Derived MSCs
  Arms: Autologous Adipose Derived MSCs
Other: Control — Standard Therapy
  Arms: Control

SUMMARY:
Despite intense research efforts and clinical trials, there is still no effective treatment that can prolong the survival of patients with IPF. Conventional therapeutic approach includes combination of corticosteroids, anti-oxidants, immunodepressants and immune modulatory anti-fibrotic agents to be discontinued 20 days before screening. The only, so far, therapeutic approach that has been proven effective in terms of prolonging patient's survival is lung transplantation. Nonetheless, not all the patients with IPF are eligible for lung transplantation; there is a significant proportion of these patients that finally succumb while waiting in a lung transplantation list. Therefore, there is critical need for more effective and reliable therapeutic modalities5. Adult Stem Cells (ASCs) seem to represent one of these. Therefore, it is conceivable to assume that adult-stem cells can be easily and safely be applied as a novel therapeutic agent in chronic and fatal lung diseases, including chronic obstructive pulmonary disease (COPD) and IPF.

Therefore, there is an urgent need to provide a safe, effective and affordable treatment option for IPF patients. New diagnostic, prognostic and therapeutic strategies need to be developed to reduce the burden of IPF. Given the present lack of appropriate treatment adjunctive in the therapy of IPF, adipose derived stromal vascular fraction provides new opportunities for development of the same.

MSCs are having anti-fibrotic activity and hence may be excellent source to tackle pulmonary fibrosis and hence could be explored for their therapeutic potential for treating Idiopathic pulmonary fibrosis. MSC's also display membrane-bound and insoluble secreted molecules involved with cell attachment to neighbouring cells and to the extra cellular matrix.18 This cell surface configuration may enable mesenchymal stem cells to home from bloodstream to mesenchymal tissue.14

As limited clinical information is available about use of SVF and MSC in the IPF patients hence this Open Label, Prospective, Randomized multi center comparative study has been undertaken to explore the tolerability & effectiveness of SVF in one treatment arm and MSC in second treatment arm in IPF patients.

Adipose derived stromal vascular fraction and Mesenchymal Stem Cells has been found in preclinical studies to be safe and effective

DETAILED DESCRIPTION:
Adipose Derived Stromal Vascular Fraction (ADSVF) Stromal Vascular Fraction (SVF) obtained from tumescent liposuction. The SVF contains a variety of cells such as pre-adipocytes, endothelial cells, smooth muscle cells, pericytes, fibroblasts, and adult stem cells (ASCs). In addition, the SVF also contains blood cells from the capillaries supplying the fat cells. These include erythrocytes or red blood cells, B and T cells, macrophages, monocytes, mast cells, natural killer (NK) cells, hematopoietic stem cells and endothelial progenitor cells, to name a few. It also contains growth factors such as transforming growth factor beta (TGF-β), platelet-derived growth factor (PDGF), and fibroblast growth factor (FGF), among others. This is consistent with the secretions of cells in the presence of an extracellular matrix. The SVF also contains the various proteins present in the adipose tissue extracellular matrix of which laminin is of interest due to its ability to help in neural regeneration.Entire procedure for SVF preparation and isolation of SVF cells will be carried out in cGMP compliance clean room.

Pure stromal vascular fraction to the tune of 99% will be isolated for this clinical trial eliminating other unnecessary cells such as RBC and leukocytes.

Adipose Derived Mesenchymal Stem Cells (ADMSC) Human mesenchymal stem cells (MSCs) are present as a rare population of cells in adipose tissue which is almost 30-40% of the nucleated cells, but they can rapidly grow in culture without losing their stemness. MSCs can be expanded in vitro ≥ 2 million -fold and retain their ability to differentiate into several mesenchymal lineages. MSCs have several characteristics such as Ease of isolation, High expansion potential,Genetic stability,Reproducible attributes from isolate to isolate,Reproducible characteristics, Compatibility with tissue engineering principles, Potential to enhance repair in many vital tissues, Uniform dose and Better quality control and release criteria.

Beside autologous use MSC can also be used for allogenic therapy. Several studies have used allo-MSC in vivo and experience suggests that the allo-MSCs are not rejected and many have positive effects on engraftment.MSC's can be isolated from various tissues, cultured ex vivo, and expanded many fold.18 Cultured-expanded MSC's appear to represent a homogeneous population by flow cytometric measures of cell-surface markers. These cell retain the ability to undergo in vitro differentiation to osteogenic, adipogenic and chondrogenic lineages, even when clonally expanded.19 Human adipose tissue derived MSCs are capable of differentiating into endothelial cells in vitro and later form capillary-like structures in semisolid medium and suggest differentiation potential of MSCs is not restricted to mesodermal lineages but also transdifferentiation of MSCs into other lineages like endothelial could be realized in vitro and in vivo8 MSCs are known to give rise to limb-bud mesoderm (osteoblasts, chondrocytes, adipocytes, stroma cells, and skeletal myoblasts) and can also differentiate into cells of visceral mesoderm (endothelial cells).9 MSCs can facilitate vasculogenesis by increasing vascular endothelial growth factor (VEGF) levels. After MSCs are intramyocardially injected into the infarct zone, local VEGF levels rise, vascular density and regional blood flow increases, and contractility improves.

MSCs are having anti-fibrotic activity and hence may be excellent source to tackle pulmonary fibrosis and hence could be explored for their therapeutic potential for treating Idiopathic pulmonary fibrosis. MSC's also display membrane-bound and insoluble secreted molecules involved with cell attachment to neighboring cells and to the extra cellular matrix.18 This cell surface configuration may enable mesenchymal stem cells to home from bloodstream to mesenchymal tissue.

ELIGIBILITY:
Inclusion:

1. Subjects aged 30 to 70 years.
2. Diagnosed subjects of IPF (HRCT scan suggestive or consistent with a probable diagnosis of usual interstitial pneumonia)
3. Diagnosis of IPF ≥ three months before enrolment in the study. In addition, the following functional abnormalities must be present:

   * Dyspnoea score of at least 2, on a scale of 0 (minimum) to 4 (maximum) on Modified Medical Research Council (MRC) scale
   * Forced Vital Capacity (FVC) of no more than 50 to 80 percent of the predicted value
   * Diffusing Lung Capacity for Carbon Monoxide (DLCO) 30 to 80 percent of the predicted value
4. The subject should be stable and able to walk ≥ 50 meters in the 6MWT. If supplemental oxygen is needed, this should not exceed 4 litres per min at rest.
5. Subjects with adequate subcutaneous fat available for liposuction as assessed by the Plastic Surgeon before liposuction procedure.
6. Subjects who have been found medically fit by the chest physician for the use sedation and/ local anesthetic before the Liposuction procedure, INR value of below 2 before liposuction procedure
7. Subject who are not currently on or have discontinued treatment with immune-suppressants and/or corticosteroids within at least 20 days prior to screening.
8. Non-pregnant, non-lactating females of age ≥18 years, and woman of childbearing potential
9. Men who are sexually active and agree to routinely use barrier method from screening and throughout the course of the study or who have undergone sterilization.

Exclusion:

1. Newly diagnosed subjects of IPF who have not received any treatment for the disease or are drug naïve subjects of IPF.
2. Subjects with a diagnosis of severe Pulmonary hypertension and a Mean Pulmonary Arterial Pressure (mPAP) of >50 mm of Hg by 2D-Echo.
3. Forced Vital Capacity (FVC) less than 50 percent of the predicted value
4. Diffusing Lung Capacity for Carbon Monoxide (DLCO) less than 30 percent of the predicted value
5. History of interstitial pulmonary fibrosis due to collagen vascular disease, connective tissue disorders and autoimmune disease
6. Subjects with any type of cancer or other serious concomitant diseases including tuberculosis, granulomatous lung disease (e.g. Sarcoidosis) or any condition in the investigator's opinion that will make the ineligible for the study
7. History of clinically significant environmental exposure, ingestion of a drug or cases of pulmonary fibrosis due to hypersensitivity pneumonitis
8. History of unstable or deteriorating cardiac or pulmonary disease other than IPF within the 6 months prior to enrolment.
9. Subjects who are pregnant, breast-feeding or have childbearing potential and have had a positive pregnancy test prior to receiving the therapy.
10. Subject who has received treatment with an investigational drug within prior 3 months or is otherwise participating in another clinical study
11. Subject who has undergone surgery within 30 days prior to screening or has planned major surgery.
12. Subject/Subject's LAR/impartial witness not willing or able to give written informed consent to participate in the study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Safety | 9 Month
  The Incidence of treatment emergent Adverse Event (AE) in the study.

SECONDARY OUTCOMES:
Efficacy | 9 Month
  Change in predicted FVC% at EOS Change in predicted DLCO% at EOS Change in the 6MWT at EOS Changes in the disease extent and severity as reflected by HRCT (64 SLICE) at EOS from randomisation.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ashok A Mahashur, M.B.B.S.M.D., Principal Investigator — P.D. Hinduja National Hospital and Medical Research Centre; Dr. Pratibha S Singhal, M.B.B.S.M.D., Principal Investigator — Bombay Hospital and Medical Research Council; Dr.Sujeet K Rajan, M.B.B.S.M.D., Principal Investigator — Bhatia General Hospital; Dr. Kartik B Shah, M.B.B.S.M.D., Principal Investigator — Cumballa Hill Hospital And Heart Institute
Locations (1):
- Kasiak Research Pvt Ltd, Thane, Maharashtra, India